CLINICAL TRIAL: NCT04712591
Title: Electrophysiologic Biomarkers of Consciousness (EBC) Recovery After Brain Injury
Brief Title: The EBC Recovery Study
Status: Recruiting | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Ayham Alkhachroum, Associate Professor of Neurology, University of Miami
Other Study IDs: 20191143
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Traumatic Brain Injury; Intracerebral Haemorrhage; Subarachnoid Haemorrhagic Stroke
Keywords: Consciousness; Coma; Recovery; Electroencephalogram
MeSH Terms: conditions — Brain Injuries, Traumatic; Cerebral Hemorrhage; Coma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute Brain Injury Patients: Acute brain injury (ABI) patients will be recruited and studied using electroencephalogram (EEG) to monitor their brain response to auditory and visual stimuli.
  Interventions: Diagnostic Test: Auditory stimuli
- Healthy Volunteers: Healthy volunteers will serve as the control group and will undergo electroencephalogram (EEG) to monitor their brain response to auditory and visual stimuli.
  Interventions: Diagnostic Test: Auditory stimuli

INTERVENTIONS:
Diagnostic Test: Auditory stimuli — Auditory stimuli (passive, active perturbations)

SUMMARY:
The purpose of this research study to find out if clinically unconscious acute brain injury patients that show brain activation to music and language on electroencephalogram (EEG) (bedside test) have better outcomes and wake up in the future.

ELIGIBILITY:
Inclusion Criteria:

For ABI Participants

* ABI adult (18 years and older) patients who are admitted to the intensive care unit
* Unconscious with Glasgow Coma Scale (GCS) <8 on presentation and unable to follow bedside commands.
* A negative COVID-19 test on arrival

For Healthy Volunteers:

* 18 years and older

Exclusion Criteria:

For All Participants:

* <18 years of age
* Pregnant woman
* Patients with cardiac arrest on presentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who present to the intensive care unit after ABI and are unconscious. Additionally, healthy volunteers will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-06-18 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Glasgow Outcome Scale-Extended (GOSE) Scale | Up to 5 years
  The GOSE is an outcome scale, range 1-8 evaluating the patients' functional outcomes - higher score indicates better recovery

SECONDARY OUTCOMES:
Coma Recovery Scale - Revised (CRS-R) | Up to 5 years
  The CRS-R will evaluate the patients' conscious state, range 0-23 -higher score indicates a better conscious state

CONTACTS AND LOCATIONS:
Overall Officials: Ayham Alkhachroum, MD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - Jackson Memorial Hospital, Miami, Florida
  - Columbia University, New York, New York

IPD SHARING:
Plan to Share IPD: No